CLINICAL TRIAL: NCT01783743
Title: Identification of TT Cases by Community Treatment Assistants: An Assessment
Acronym: SIMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Lions Club International Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NA_00043444
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-02

CONDITIONS: Trichiasis
Keywords: Trichiasis; Trachoma; Mass treatment
MeSH Terms: conditions — Trichiasis; Trachoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): Community treatment assistants (CTA ) will receive usual training, including the basic background of trachoma/trichiasis recognition, drug administration, and azithromycin dosing.
  In addition to the usual training, these CTA's will also receive an additional modest half day training for TT case recognition which is called the TT training program and TT Screening Card to help them identify TT cases and refer them for surgery.
  Interventions: Other: TT Training Program and TT Screening Card
- Usual Assessment arm (No Intervention): Community treatment assistants will receive only usual training, including the basic background of trachoma/trichiasis recognition, drug administration, and azithromycin dosing.

INTERVENTIONS:
Other: TT Training Program and TT Screening Card — The intervention is an additional half day training program on trichiasis recognition (TT Training Program) and a TT Screening card to assist community treatment assistants in recognizing TT cases and referring them to surgery.
  Arms: Intervention arm

SUMMARY:
To achieve the goal of trachoma control as mandated by the World Health Organization, countries must reduce the backlog of trichiasis surgery cases to less than 1/1,000 of their population. However, these cases reside in rural villages in trachoma endemic districts, and finding them to offer services is a challenge. Community Treatment Assistants (CTAs) are village residents who are trained to offer Mass Drug Administration (MDA) to their communities and hence are in contact with most residents. A training guide and tool for screening for trachomatous trichiasis (TT) will be developed to train CTAs in rural Tanzania to identify cases in their communities and refer them to surgery. Compared to the current process by which CTAs passively screen for TT if cases complaint, investigators hypothesize that the trained CTAs will identify twice the usual number of TT surgery cases during ongoing community antibiotic administrations for trachoma and will also miss fewer cases. If this simple system is effective, it can be implemented widely to screen communities for cases of TT.

Residents from thirty-six villages holding MDA, for whom a complete census is available, will be randomized on a 1:1 basis to intervention (where the CTAs receive the enhanced training from the enhanced training team) and usual assessment (where the CTAs receive the usual instructions from the regular MDA team). In both arms, the CTAs will keep records of all cases they have screened as positive for TT amongst the residents.

A Master TT grader will grade all screened cases of TT to determine the rate of true positivity in both arms.In addition, he will examine a random sample of residents who are screened as negative to detect potentially missed cases and estimate the total burden of trichiasis cases in both arms as well.The assessments of the Master TT grader will serve as the gold standard for calculations of sensitivity, specificity, and positive and negative predictive values of the enhanced training versus usual assessment methods.

ELIGIBILITY:
Inclusion Criteria:

* All persons in the study and control communities are eligible for the MDA.
* Adults aged 15 and over will be eligible for the survey and re-assessment.
* Those who are screened positive in the re-assessment will be eligible for treatment at the surgery camp.
* Those who are screened positive for TT initially but refuse the definitive re-screening will still be offered surgery but told they may not have TT and will be re-screened by the surgeon.

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27473 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K West, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community randomized trial was conducted in 36 communities during MDA .Community served as unit of randomization & enrolled villages were randomly allocated on 1:1 basis to either intervention (n=18) or usual care (n=18) arms.Total MDA eligible population in control arm was 13509 individuals and in the intervention arm was 13964 individuals.
Pre-assignment Details: Community Treatment Assistants(CTAs) in intervention arm received an additional half-day training and TT screening card in addition to training received by CTAs in usual care arm. All MDA participants 15 years and older were screened for TT.Senior grader re-screened all TT cases identified by CTAs along with a selected random sample in both arms.
Units Other Than Participants: communities
Groups:
- Control (Usual Assessment): Community treatment assistants will receive usual training, including basic background of trachoma/trichiasis recognition, drug administration and azithromycin dosing.
- Intervention (Novel TT Screening Tool): Community treatment assistants will receive usual training, including basic background of trachoma/trichiasis recognition, drug administration and azithromycin dosing, plus a modest additional TT Training Program and Recognition Card.
  TT Training Program and Recognition Card: The intervention is an additional training program on trichiasis recognition and a TT recognition card to assist community treatment assistants in recognizing TT cases and referring them to surgery.
Period: Screening of Subjects by CTA During MDA
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Started | 13509; 18 communities | 13964; 18 communities
Completed | 10082; 18 communities | 9525; 18 communities
Not Completed | 3427; 0 communities | 4439; 0 communities
Not completed — Absent at MDA | 3427 | 4439
Period: Rescreening of Subjects by Senior Grader
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Started | 13509; 18 communities | 13964; 18 communities
TT Positive Cases Screened by CTA | 46; 18 communities | 409; 18 communities
Random Sample From Non TT Cases by CTA | 1721; 18 communities | 1786; 18 communities
Random Sample From Subject Absent at MDA | 846; 18 communities | 849; 18 communities
Completed | 2613; 18 communities | 3044; 18 communities
Not Completed | 10896; 0 communities | 10920; 0 communities
Not completed — Lost to Follow-up | 591 | 684
Not completed — Not part of the random sample selected | 10305 | 10236

BASELINE CHARACTERISTICS:
Units Other Than Participants: community
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool) | Total
Number analyzed (Participants) | 13509 | 13964 | 27473
Number analyzed (community) | 18 | 18 | 36
Age, Customized [Median (Inter-Quartile Range); unit: participants]
  15-39 years | 494 [327 to 682] | 482 [398 to 644] | 488 [364 to 663]
  40-59 years | 168 [97 to 203] | 152 [119 to 206] | 160 [108 to 205]
  60 and older | 81 [54 to 107] | 83 [67 to 108] | 82 [61 to 108]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7160 | 7401 | 14561
  Male | 6349 | 6563 | 12912
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 13509 | 13964 | 27473

OUTCOME MEASURES:

1. Primary Outcome: TT Cases Screened Positive by CTA's and Confirmed by Graders
Description: All the TT cases detected in control versus intervention arms (adjusted for population size) through screening were verified by graders.
  Grader re-graded all these cases except for the cases lost to follow-up.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Number analyzed (Participants) | 32 | 316
Participants | 9 | 50

2. Secondary Outcome: Sensitivity of TT Screening Methods
Description: Sensitivity of different TT screening methods compared to "true" assessment of cases and controls using the extrapolated values from the follow-up survey.
  Formula used: True positives/(true positives +false negative)
Time Frame: 10 months
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Number analyzed (Participants) | 46 | 409
percentage of true positives | 5.7 [2.6 to 8.6] | 31.2 [24.9 to 37.6]

3. Secondary Outcome: Specificity of TT Screening Methods
Description: Specificity of different TT screening methods compared to "true" assessment of cases and controls using the extrapolated values from the follow-up survey.
  Formula used: True negatives/(true negatives +false positive)
Time Frame: 10 months
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Number analyzed (Participants) | 10036 | 9116
percentage of true negatives | 99.7 [99.6 to 99.8] | 98.0 [97.6 to 98.2]

4. Secondary Outcome: Positive Predictive Values of TT Screening Methods
Description: Positive Predictive Values (PPV) of the different screening methods compared to "true" assessment of cases and controls.
  It was calculated by using extrapolated values. The formula used: True positives /total participants at initial screening screened as positive by CTA's.
Time Frame: 10 months
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Number analyzed (Participants) | 46 | 409
percentage of true positives | 28.1 [15.1 to 41.1] | 15.8 [12.3 to 19.4]

5. Secondary Outcome: Negative Predictive Values of TT Screening Methods
Description: Negative Predictive Values (NPV) of the different screening methods compared to "true" assessment of cases and controls.
  It was calculated by using extrapolated values. Formula used : True Negatives /total participants at initial screening,screened as negative by CTA's
Time Frame: 10 months
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Number analyzed (Participants) | 10036 | 9116
percentage of true negatives | 98.0 [97.6 to 98.2] | 2.2 [2.0 to 2.5]

ADVERSE EVENTS:
Time Frame: 10 months (Between January 2013 to November 2013)
Arm/Group | Control (Usual Assessment) | Intervention (Novel TT Screening Tool)
Serious Adverse Events (participants affected / at risk) | 0/13509 | 0/13964
Other Adverse Events (participants affected / at risk) | 0/13509 | 0/13964

LIMITATIONS AND CAVEATS:
1. While use of CTAs in TT screening during MDA offers clear advantages, this approach is limited to areas that merit MDA.
2. Attrition of CTAs may also prove to be a limitation for this screening approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes